CLINICAL TRIAL: NCT06872372
Title: Role of N-Acetylcysteine in Non-Acetaminophen-Induced Acute Liver Failure: a Randomized Controlled Trial
Brief Title: Role of N-Acetylcysteine in Non-Acetaminophen-Induced Acute Liver Failure
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore General Hospital (Other Government)
Responsible Party: Principal Investigator, Muhammad Irfan Jamil, Principal Investigator, Lahore General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LahoreGeneralH3
Record Dates: First submitted 2025-02-27; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Acute Liver Failure; Drug-Induced Liver Injury
Keywords: Non-Acetaminophen-Induced Liver Injury; N-Acetylcysteine (NAC); Drug-Induced Hepatotoxicity
MeSH Terms: conditions — Liver Failure, Acute; Chemical and Drug Induced Liver Injury | interventions — Acetylcysteine; Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NAC Group (Experimental): Participants in this group received N-Acetylcysteine (NAC) along with standard supportive care for acute liver failure. NAC was administered orally or via a nasogastric tube.
  Interventions: Drug: N-Acetylcysteine (NAC) Treatment
- Control Group (Placebo Comparator): Participants in this group received only standard supportive care, without N-Acetylcysteine (NAC).
  Interventions: Other: Standard supportive care

INTERVENTIONS:
Drug: N-Acetylcysteine (NAC) Treatment — Participants in this group received N-Acetylcysteine (NAC) at a dose of 140 mg/kg orally or via a nasogastric tube every 4 hours for the first 16 hours, followed by the same dose at intervals of 6-8 hours for a total of 3 days, alongside standard supportive care for acute liver failure.
  Arms: NAC Group
Other: Standard supportive care — Participants in this group received only standard supportive care for acute liver failure, without N-Acetylcysteine (NAC). Standard supportive care included measures to prevent hypoglycemia, administration of broad-spectrum antimicrobials, proton pump inhibitors, fluid and electrolyte balance maintenance, and supportive treatment for hepatic encephalopathy.
  Arms: Control Group

SUMMARY:
Acute liver failure (ALF) is a serious condition in which the liver suddenly stops working, often leading to life-threatening complications. While N-Acetylcysteine (NAC) is widely used to treat ALF caused by acetaminophen overdose, its benefits in ALF due to other causes, such as viral infections or drug reactions, remain uncertain.

This study is a randomized controlled trial designed to investigate whether NAC can improve survival rates and reduce hospital stays in patients with non-acetaminophen-induced ALF. Participants will be randomly assigned to receive either NAC along with standard supportive care or standard supportive care alone. The study will measure survival rates, hospital stay duration, and improvement in liver function tests.

By exploring NAC's potential benefits beyond acetaminophen-related cases, this research aims to provide evidence-based guidance on how to better manage patients with ALF from other causes.

DETAILED DESCRIPTION:
This study was conducted with the necessary ethical considerations. Ethical approval was obtained from the ethical review board of the institution. Informed consent was obtained from each participant or their legal guardians before enrollment in the study. Participants were selected based on predefined selection criteria. Comprehensive baseline data were gathered from all participants, including demographic information (age, gender), detailed medical history (duration of symptoms, known etiologies), and past medical conditions (comorbidities, chronic viral hepatitis, tuberculosis).

Baseline investigations included a comprehensive set of laboratory tests: bilirubin, albumin, International Normalized Ratio (INR), Aspartate Aminotransferase, Alanine Aminotransferase, complete blood count, renal function tests, electrolytes, blood glucose, and viral serology (Hepatitis B Surface Antigen, Hepatitis B Core Immunoglobulin M, Hepatitis A Virus Immunoglobulin M, Hepatitis C Virus Antibody), along with additional tests as indicated by clinical suspicion (e.g., autoimmune markers, Wilson profile, iron profile, Herpes Simplex Virus / Cytomegalovirus / Epstein-Barr Virus serology). All patients were admitted to the Intensive Care Unit. Participants were randomly assigned to either the NAC treatment group or the control group using the lottery method.

NAC Group: NAC was administered at a dose of 140 mg/kg orally or via a nasogastric tube every 4 hours for the first 16 hours, followed by the same dose at intervals of 6-8 hours. It was continued for 3 days.

Control Group: Participants received the standard supportive care protocol for ALF.

Throughout the study, participants received standard supportive care treatment, which remained consistent in both groups. This care included measures to prevent hypoglycemia, the administration of broad-spectrum prophylactic antimicrobials, proton pump inhibitors for stress-related ulcers, and maintenance of fluid and electrolyte balance. In cases of advanced hepatic encephalopathy, anti-encephalopathy measures were provided. Fresh frozen plasma was administered to patients experiencing spontaneous bleeding. Blood and urine cultures were obtained in cases where sepsis was suspected, and treatment was administered based on sensitivity. Patients were followed for up to 28 days to assess outcomes. Data were collected using a data collection proforma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with either gender (male or female) aged 18-60 years.
* Diagnosed with non-acetaminophen-induced acute hepatic failure (NAI-AHF) as per operational definition.
* Cases where the etiology is attributed to factors other than acetaminophen overdose, including viral hepatitis (HAV, HBV, HEV), drug-induced liver injury (excluding acetaminophen), or idiopathic causes.
* Patients who have not received N-acetylcysteine (NAC) treatment for the current episode of acute hepatic failure before enrollment.

Exclusion Criteria:

* Patients with a history of chronic liver disease or cirrhosis.
* Patients with previous history of severe cardiac, renal, neurological, or infectious diseases that could confound treatment outcomes.
* Patients who have undergone a liver transplant or potential candidate of liver transplant.
* Known allergy or contraindication to N-acetylcysteine.
* Pregnant women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Survival Rate | 28 days post-enrollment
  It is defined as the proportion of patients with non-acetaminophen-induced acute liver injury who remain alive at 28th day after enrollment.
Mortality Rate | 28 days post-enrollment
  Proportion of patients who die within 28 days after enrollment in the study.

SECONDARY OUTCOMES:
Length of Hospital Stay | Through study completion, an average of 28 days
  The total number of days each participant hospitalized from admission to discharge or death.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Irfan Jamil, Principal Investigator — Lahore General Hospital, Lahore
Locations (1):
- Lahore General Hospital, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No